CLINICAL TRIAL: NCT04243837
Title: A Phase 2a Double-Blind, Placebo-Controlled Study to Determine the Safety, Tolerability, Pharmacokinetics, and Efficacy of Deupirfenidone (LYT-100) in Patients With Breast Cancer-Related Upper Limb Secondary Lymphoedema
Brief Title: LYT-100 in Patients With BCRL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary objective/endpoint has been established, will not pursue development of the disease indication further
Sponsor: PureTech (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LYT-100-2020-US-02
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer Related Lymphoedema; Lymphoedema
MeSH Terms: conditions — Lymphedema | interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: Consists of 1 cohort with 2 arms: active treatment or placebo patients
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LYT-100 in patients with BCRL (Experimental): LYT-100 BID for 6 months
  Interventions: Drug: LYT-100 BCRL
- Placebo in patients with BCRL (Placebo Comparator): Placebo BID for 6 months
  Interventions: Drug: Placebo BCRL

INTERVENTIONS:
Drug: LYT-100 BCRL — BCRL patients will receive LYT-100 BID for 6 months
  Other Names: Deupirfenidone
  Arms: LYT-100 in patients with BCRL
Drug: Placebo BCRL — BCRL patients will receive Placebo BID for 6 months
  Other Names: Placebo
  Arms: Placebo in patients with BCRL

SUMMARY:
This is a trial of up to 6-months duration for safety, tolerability, clinical efficacy assessments, PK and biomarkers analysis in breast carcinoma patients with secondary lymphoedema

DETAILED DESCRIPTION:
This trial will utilize a randomised, double-blinded, placebo controlled design that will assess the safety, tolerability, and secondarily clinical efficacy of LYT-100 over a period of up to 6-months of dosing in breast carcinoma patients with secondary lymphoedema following sentinel lymph node biopsy and/or axillary node dissection, with or without radiation.

ELIGIBILITY:
Main Inclusion Criteria:

1. Female or male between 18 and 80 years old (inclusive) at the time of informed consent.
2. At least 6 months since any type of breast cancer surgery (excluding fine needle aspiration biopsy [FNA]), at the time of study screening. No intention to have breast reconstructive surgery, nipple reconstruction and/or tattooing during the course of the study.
3. At least 3 months since completion of all types of treatment for breast cancer, including but not limited to neoadjuvant, radiotherapy, chemotherapy and immunotherapy, at the time of study screening.
4. At least 3 months treatment of stable adjuvant treatment with hormonal or anti-HER2 therapy at the time of screening, with no planned changes to this therapy throughout the duration of the study.
5. Diagnosis of primary breast cancer, and without evidence of recurrence of breast cancer and/or metastasis for at least 6 months since breast cancer surgery, as determined at screening and baseline.
6. Documented evidence of Stage 1 or 2 lymphedema.
7. Receiving standard of care compression or agreeable to using care compression, or no compression at all ≥ 4 weeks prior to screening and throughout the study.

Main Exclusion Criteria:

1. Bilateral lymphoedema or history of bilateral axillary lymph node removal (i.e., sentinel lymph node or axillary lymph node dissection), or primary lymphoedema or lymphatic or vascular malformation, determined at screening.
2. Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within 3 months prior to study drug administration; corticosteroids are permitted at the discretion of the PI.
3. Recent history (in the 8 weeks prior to screening) of cellulitis, lymphangitis, dermatitis, necrotizing fasciitis, or current open wounds or sores in the affected extremity.
4. Stage III lymphoedema, or history of clinically diagnosed secondary lymphoedema greater than 4 years, determined at screening.
5. Initiated use of compression or manual lymphatic drainage or other lymphoedema therapies at the start of the study within 4 weeks of the screening visit. Rescreening is allowed following a course of stable compression regimen of > 4 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - MACRO Trials, Los Angeles, California
  - Accel Research Network, Maitland, Florida
  - Accel Research Network, Atlanta, Georgia
- Australia (4):
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - Ballarat Health Services, Ballarat, Victoria
  - Flinders University, Adelaide
  - Macquarie University Health Sciences Centre, Sydney

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen MC, Korth CC, Harnett MD, Elenko E, Lickliter JD. A Randomized Phase 1 Evaluation of Deupirfenidone, a Novel Deuterium-Containing Drug Candidate for Interstitial Lung Disease and Other Inflammatory and Fibrotic Diseases. Clin Pharmacol Drug Dev. 2022 Feb;11(2):220-234. doi: 10.1002/cpdd.1040. Epub 2021 Nov 15. PMID 34779583

RESULTS

PARTICIPANT FLOW:
Groups:
- LYT-100 in Patients With BCRL: LYT-100 BID for 6 months
  LYT-100 BCRL: BCRL patients will receive LYT-100 500 mg BIDX3 days followed by LYT-100 750 mg BID for 6 months
Period: Overall Study
Arm/Group | LYT-100 in Patients With BCRL | Placebo in Patients With BCRL
Started | 28 | 22
Completed | 10 | 7
Not Completed | 18 | 15
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Covid-19 lock down | 1 | 0
Not completed — Study Terminated by Sponsor | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- LYT-100 in Patients With BCRL: LYT-100 BID for 6 months
  LYT-100 BCRL: BCRL patients will receive LYT-100 500mg BID x3 days followed by LYT-100 750mg BID for 6 months
- Total: Total of all reporting groups
Arm/Group | LYT-100 in Patients With BCRL | Placebo in Patients With BCRL | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 7 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 28 | 20 | 48
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
  Australia | 19 | 13 | 32

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Evaluate the safety and tolerability of LYT-100 as measured by TEAEs
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | LYT-100 in Patients With BCRL | Placebo in Patients With BCRL
Number analyzed (Participants) | 28 | 22
Participants | 22 | 13

ADVERSE EVENTS:
Time Frame: 6 months
Description: Systemic Assessment methods were used to routinely evaluate if any adverse events have occurred. Examples of these methods include: regular investigator assessments through physical exams and laboratory testing.
Arm/Group | LYT-100 in Patients With BCRL | Placebo in Patients With BCRL
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/28 | 2/22
Other Adverse Events (participants affected / at risk) | 22/28 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYT-100 in Patients With BCRL (N=28) | Placebo in Patients With BCRL (N=22)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LYT-100 in Patients With BCRL (N=28) | Placebo in Patients With BCRL (N=22)
Nausea (Gastrointestinal disorders) | 13 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 0
COVID-19 (Infections and infestations) | 4 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2
Headache (Nervous system disorders) | 4 | 3
Dizziness (Nervous system disorders) | 0 | 2
Fatigue (General disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04243837/Prot_SAP_001.pdf